CLINICAL TRIAL: NCT05296642
Title: Exploring the Use of Blood Flow Restriction in Addition to Aerobic Exercise as a Modality to Produce Exercise Induced Hypoalgesia in Participants With Painful Diabetic Peripheral Neuropathy.
Brief Title: Exercise Induced Hypoalgesia Diabetes
Acronym: EIHDM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator decision
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Marlon Wong, Assistant Professor, University of Miami
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 20220189
Record Dates: First submitted 2022-03-16; First posted 2022-03-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Diabetic Peripheral Neuropathy; Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cycling at a Moderate Intensity Aerobic Exercise (AE) group (Experimental): All participants will be asked to cycle during the first phase at a moderate intensity for 20 minutes.
  Interventions: Other: Moderate Cycling
- Blood Flow restriction training with cycling at a moderate intensity (BFR+AE) group (Experimental): All participants will be asked to wear an automated personalize tourniquet system to restrict blood flow. Participants will be asked to lie in supine and a non-shedding stockinette protection sleeve will be placed at bilateral proximal thighs. Then, participants will be asked to cycle at a moderate intensity for 20 minutes during the second phase.
  Interventions: Other: Moderate Cycling; Other: Personalized Tourniquet System

INTERVENTIONS:
Other: Moderate Cycling — Using the recumbent bicycle (95Ri, Life Fitness, Illinois) participants will be asked to sustain a moderate pace of 13 - 16 for 20 minutes of perceived exertion range using the Borg rate of perceived exertion scale (RPE).
Other: Personalized Tourniquet System — An automated personalize tourniquet system (Delfi Medical, Inc., Vancouver, BC, Canada) will be used to perform blood flow restriction during BFR+AE. This system has a dual-purpose tourniquet cuff (11.5 x 86 cm) connected by airtight hose tubing to a personalized tourniquet device. The device automatically measures LOP and regulated pressure during exercise within clinically acceptable limits. Participants will be asked to lie in supine and a non-shedding stockinette protection sleeve will be placed at bilateral proximal thighs. Following, a tourniquet cuff will be placed bilaterally around the protection material and connected to the airtight hose tube.
  Arms: Blood Flow restriction training with cycling at a moderate intensity (BFR+AE) group

SUMMARY:
The purpose of this research study is to learn whether different forms of exercise can reduce pain experienced by individuals with painful diabetic peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 18 - 65.
2. Subjects with confirmed Diabetes Mellitus as defined by the American Diabetes Association (ADA), a glycosylated hemoglobin (HbA1c) of 6.5%, a fasting blood glucose > 126 mg/dL, or an oral glucose tolerance test > 200 mg/dL.
3. Subjects who have stocking and/or glove distribution neuropathy symptoms as drawn on the painDETECT questionnaire.
4. Subjects who have neuropathic pain as defined by a minimum score of 4 or higher on the Douleur Neuropathique en 4 Questions (DN4). In addition, the location of pain must be present within the same region of neuropathy symptoms.
5. Subjects who have an ankle brachial index (ABI) between 0.7 and 1.4.

Exclusion Criteria:

1. Subjects who have pain due to some other form of neuropathy (chemo-induced neuropathy, alcohol induced neuropathy, exposure to toxins/chemicals, vitamin b12 deficiency, etc.) assessed via a medical history.
2. Subjects with current or history of central nervous system disorders.
3. Subjects with resting hypertension (HTN) >/= 160/90 mmHg or known uncontrolled hypertension, coronary artery disease, heart failure, retinopathy, chronic obstructive pulmonary disease, end-stage renal disease, or current open foot ulcers.
4. Subjects who are unable to achieve walking a minimum distance of 400 meters in the six-minute walk test.
5. Subjects with Reynaud's disease or cold urticaria.
6. All vulnerable populations including adults unable to consent, individuals who are not yet adults (infants, children, teenagers), pregnant women, prisoners, individuals with cognitive impairment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Pressure Threshold (PPT) | Baseline, 20 minutes
  PPT will be measured both locally at the quadriceps and distally at the upper trapezius. The PPT will be determined with three series of ascending stimulus intensities at each point over 3 rounds. A positive change in PPT (PPT following exercise subtracted from PPT before exercise) will demonstrate an intact exercise induced hypoalgesic response.

SECONDARY OUTCOMES:
Change in Heat Pain Threshold (HPT) | Baseline, 20 minutes
  HPT will be measured both locally at the quadriceps and distally at the upper trapezius. The HPT will be determined with three series of ascending stimulus intensities at each point over 3 rounds. A positive change in HPT (HPT following exercise subtracted from HPT before exercise) will demonstrate an intact exercise induced hypoalgesic response.

CONTACTS AND LOCATIONS:
Overall Officials: Marlon L. Wong, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No